CLINICAL TRIAL: NCT03115541
Title: The Contemporary Significance of Deep Venous Thrombosis and Pulmonary Embolus in Patients Undergoing Esophagectomy: A Pilot Study to Evaluate the Incidence of DVT and PE After Major Esophageal Resections
Brief Title: Incidence of Venous Thromboembolism in Patients Undergoing Major Esophageal Resection
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: SJHH_VTEesoph001
Record Dates: First submitted 2017-02-22; First posted 2017-04-14 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Venous Thromboembolism; Thoracic Surgery; Esophageal Cancer
Keywords: venous thromboembolism prophylaxis; deep vein thrombosis; pulmonary embolus; esophageal resection; incidence
MeSH Terms: conditions — Venous Thromboembolism; Esophageal Neoplasms; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the incidence of post-operative venous thromboembolism (VTE) in patients undergoing major esophageal resection for malignancy.

DETAILED DESCRIPTION:
Venous Thromboembolism (VTE) is a common post-operative complication that can result in significant patient morbidity, mortality and health care resource utilization to treat the resultant Pulmonary Embolus (PE) or Deep Vein Thrombosis (DVT) events. It is the third leading cause of cardiovascular mortality. Due to the high burden of disease, VTE events are actively prevented using mechanical and/or pharmaceutical prophylaxis interventions such as compression stockings or a variety of anti-coagulants. Extensive literature identifies incidence rates and provides guidelines regarding the use of prophylaxis measures in orthopaedic and oncological surgery, but the literature in thoracic surgery is sparse at best or conflicting with reported incidence of symptomatic events ranging from 5% to 14% after esophagectomy. The current practice of VTE prophylaxis in thoracic surgery includes administration of unfractionated or low molecular weight heparin (LMWH) starting in the perioperative period and finishing at patient discharge, while prolonged thromboprophylaxis in orthopaedic surgery beyond 10 to 14 days and up to 35 days has become the standard of care. Such an approach has never been tested or validated in esophageal cancer patients despite the substantial burden and high risk of VTE events in this population. There is a clear need for well-designed studies aiming to define the extent of peri-operative VTE for esophagectomy patients and additional contributing factors associated with VTE in those high risk patients in order to inform best practice patterns. The investigators hypothesize that the incidence and clinical burden of perioperative VTE events in esophagectomy patients are substantial, and that VTE significantly contributes to peri-and post-operative morbidity and mortality. Hence, it will be beneficial to explore the true incidence of VTE events and evaluate the effectiveness of extended-duration, post-discharge prophylaxis for these patients. The investigators also hypothesize that sub-groups of esophagectomy patients will be at higher risk for VTE events and therefore might benefit more from extended-duration, post-discharge prophylaxis, and perhaps from a more aggressive in-hospital regimen.

This prospective cohort study will involve patients undergoing major esophageal resection for esophageal cancer at 9 tertiary care centres across Canada, 4 centres in the USA, and 1 site in China. McMaster University at St. Joseph's Healthcare Hamilton will serve as the Coordinating Centre as well as a study site. Recruitment will commence at each site until 177 patients are enrolled via consecutive convenience sampling. After undergoing esophagectomy, all patients will receive both a peri-operative dose followed by post-operative LMWH VTE prophylaxis for the remainder of their hospital stay. As per current VTE prophylaxis guidelines, prophylaxis will be discontinued upon hospital discharge. VTE outcomes will be assessed using Computed Tomography with pulmonary angiography protocol at 30 and 90 days and bilateral venous Doppler ultrasounds at 30, 60 and 90 days after surgery. The role of D-Dimer will be investigated peri-operatively up to post-operative day (POD) 3, at hospital discharge or POD 10 (whichever is applicable), and at each imaging follow-up visit. A future second phase study will be a randomized controlled trial that will evaluate the role of extended duration thromboprophylaxis post-discharge in reducing the incidence of VTE in this patient population. The proposed prospective cohort study to evaluate the incidence of VTE needs to be conducted first, in order to optimize patient selection and determine the sample size for the subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age.
2. Patients may be of either gender.
3. Patients must be diagnosed with resectable esophageal cancer.
4. Patients must be undergoing an esophagectomy as either the first-line treatment or after completion of neoadjuvant therapies.
5. Patients must receive VTE prophylaxis as per local institutional guidelines
6. Patients must be competent to understand and sign consent documents.

Exclusion Criteria:

1. All patients with known allergic or anaphylactic reaction to contrast dye, heparin, or low molecular weight heparin (LMWH).
2. Patients must not be under current anticoagulation for venous thromboembolism or other medical conditions.
3. Patients must not have known renal impairment, defined as creatinine clearance value of less than 55ml/min/m2 as calculated by the Cockcroft-Gault method.
4. Patients with a history of, or ongoing liver disease, manifested as ascites or previous peritoneal tapping for ascites.
5. Patients with known hepatic insufficiency, defined as international normalized ratio (INR) >1.5.
6. Patients must not be pregnant or planning to become pregnant.
7. Patients must not have been diagnosed or treated for VTE in the past 3 months prior to surgery.
8. Patients must not have a present or previous increased risk of haemorrhage.
9. Patients must not have known, objectively confirmed bleeding and clotting disorders such as thrombophilia, von Willebrand's disease, hemophilia or otherwise active bleeding.
10. Patients must not have a history of previous heparin-induced thrombocytopenia (HIT).
11. Platelet count must be above 75,000, but transient, recovered thrombocytopenia associated with chemotherapy will not be a basis for exclusion.
12. Patients must not have previously inserted inferior vena cava (IVC) filter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve patients undergoing esophageal resection for malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of PE/DVT after esophageal resection for malignancies | post-operative 30 days
  CT pulmonary angiogram and bilateral leg Doppler ultrasound to assess evidence of PE/DVT
Incidence of PE/DVT after esophageal resection for malignancies | post-operative 60 days
  CT pulmonary angiogram and bilateral leg Doppler ultrasound to assess evidence of PE/DVT
Incidence of PE/DVT after esophageal resection for malignancies | post-operative 90 days
  CT pulmonary angiogram and bilateral leg Doppler ultrasound to assess evidence of PE/DVT

SECONDARY OUTCOMES:
Incidence of PE and DVT comparing open esophagectomy with minimally invasive surgery | post-operative 30, 60, 90 days
  CT pulmonary angiogram and bilateral leg Doppler ultrasound to assess evidence of PE/DVT
Complications and mortality of DVT and PE post esophageal resection | post-operative 30, 60, 90 days
  Multiple measurements aggregated to arrive at one reported value (e.g., number of participants with adverse events that are related to DVT and PE).
Risk factors for the development of VTE post esophageal resection | post-operative 30, 60, 90 days
  Multiple measurements used including patient characteristics, surgical details, physiological parameters, and patient-reported symptoms questionnaire.
Correlation between D-Dimer levels and VTE events post esophagectomy | post-operatively up to 3 days after surgery, at hospital discharge/post-operative day 10, and at 30, 60, 90 days after surgery
  Blood samples used to assess D-Dimer levels to investigate the role of this laboratory test as a quantifiable clinical measure of VTE risk.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, Principal Investigator — McMaster University
Locations (9):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
- Canada (5):
  - University of Manitoba, Winnipeg, Manitoba
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Beijing Chao-yang Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Martino RR, Goodney PP, Spangler EL, Wallaert JB, Corriere MA, Rzucidlo EM, Walsh DB, Stone DH. Variation in thromboembolic complications among patients undergoing commonly performed cancer operations. J Vasc Surg. 2012 Apr;55(4):1035-1040.e4. doi: 10.1016/j.jvs.2011.10.129. Epub 2012 Mar 10. PMID 22409858
- [Background] Mukherjee D, Lidor AO, Chu KM, Gearhart SL, Haut ER, Chang DC. Postoperative venous thromboembolism rates vary significantly after different types of major abdominal operations. J Gastrointest Surg. 2008 Nov;12(11):2015-22. doi: 10.1007/s11605-008-0600-1. Epub 2008 Jul 31. PMID 18668299